CLINICAL TRIAL: NCT01192685
Title: Transcranial Magnetic Stimulation in Major Depression With EEG and NIRS Monitoring
Brief Title: Transcranial Magnetic Stimulation in Major Depression With EEG and Near Infrared Spectroscopy (NIRS) Monitoring
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Neuronavigation system equipment failure caused unreliable data
Sponsor: Boston University (Other)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H-29098
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Depression; Depressed; TMS; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depression; Consciousness Disorders | interventions — Transcranial Magnetic Stimulation; Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Depressed outpatients treated with TMS (Other): This a 12- week study (1-4 week screening, 6 weeks treatment, 2 weeks follow-up) outpatient open label clinical trial. Twenty-five subjects diagnosed with depression with a Montgomery Asberg Depression Rating Scale (MADRAS) score of 26 or higher, will be enrolled into this trial, up to fifty subjects will be consented. Transcranial Magnetic Stimulation (TMS) will be administered to subjects 5 days a week for 6 weeks. Near infrared spectroscopy (NIRS), a spectroscopic method that uses the near infrared region of the electromagnetic spectrum (from about 700 nm to 2500 nm), will be used to assess blood flow in the brain.
  Interventions: Procedure: Transcranial Magnetic Stimulation (TMS); Device: near infrared spectroscopy (NIRS)

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation (TMS) — TMS will be administered to subjects 5 days a week-typically Monday through Friday, for 6 weeks.
Device: near infrared spectroscopy (NIRS) — near infrared spectroscopy (NIRS) will be used to measure the blood flow in the brain

SUMMARY:
This a 12- week study (1-4 week screening, 6 weeks treatment, 2 weeks follow-up) outpatient open label clinical trial. Twenty-five subjects diagnosed with depression with a Montgomery Asberg Depression Rating Scale (MADRAS) score of 26 or higher, will be enrolled into this trial, up to fifty subjects will be consented. The primary purpose of the current study is to determine: 1) if changes in electrical activity of the brain measured by EEG in specific areas is associated with changes in the blood flow of the brain 2) Which areas of the brain show changes in electrical activity and treatment response.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) has demonstrated efficacy as a treatment for major depression. No objective markers have been identified that indicate which patients are most likely to respond to TMS therapy. The goal of the present investigation is to determine whether an electroencephalographic measure called cordance or a measure of blood flow in the frontal brain, as measured by near infrared spectroscopy (NIRS) can serve as predictors of outcome with TMS therapy in depression. Subjects with depression will be treated in this study for 6 weeks with TMS. Frontal brain blood flow measured using NIRS will be assessed prior to TMS therapy, and repeatedly thereafter. EEG cordance will also be obtained following a similar schedule. Measures of depression and other psychiatric disorders will be collected prior to, during and for 2 weeks after the completion of TMS treatment. The correlation between these measures and the EEG and NIRS measures will then be determined to see if these latter measures are predictive of improvement in depression.

ELIGIBILITY:
Inclusion criteria List

1. Depressive disorder Diagnostic Statistical Manual of Mental Disorders, fourth Edition, Text Revision (DSM-IV-TR).
2. MADRAS score of 26 or above and history of depression, as defined by meeting DSM-IV criteria for major depression, dysthymic disorder, or substance-induced mood disorder.
3. Male or female aged 18 to 65.
4. Females who are not pregnant or nursing.
5. Individuals able to provide informed written consent and are able to comply with study procedures.
6. Subjects who have received or are receiving anti-depressant medication.
7. Patients who are depressed as assessed by the above criteria and have not had optimum response to their antidepressant medication in their current episode.

Exclusion criteria List

1. Any Axis I diagnosis that, in the opinion of the investigators, may interfere with the course of the trial.
2. Any current diagnoses of alcohol abuse or dependence.
3. Any current substance use disorder.
4. Medical or neurological illness that in the investigators judgment would make study compliance difficult or would be a contraindication for use with TMS.
5. Currently receiving any medication that markedly increases the risks for seizures, for example: tricyclic antidepressants, INH, meperidine, lidocaine, and clozapine.
6. Subjects who have implanted metallic devices or non-removable metallic objects in or around the head that can be magnetized, however metal fillings, braces, and dental implants are acceptable.
7. Subjects who have implanted devices that emit physiological signals including cardioverter defibrillators (ICDs), and vagus nerve stimulators.
8. Subjects who have received any investigational drug during the prior 30 days.
9. Clinically significant abnormal lab values as assesses by the Investigator.
10. Risk for suicidal behavior based on clinician assessment and a score of greater than 5 on the suicidal thought item of the MADRS or a score of 4 on the suicide item of the Hamilton Depression rating scale.
11. Subjects who have had a serious suicide attempt in the past year as assessed by the Investigator.
12. Current other somatic antidepressant therapy, i.e. vagus nerve stimulation, electroconvulsive therapy, or phototherapy.
13. Started psychotherapy in the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The correlations between EEG cordance or task-induced changes in frontal total Hb levels | 6 weeks
  The primary outcome will be the correlations between EEG cordance or task-induced changes in frontal total Hb levels and changes in MADRAS scores between baseline and the last treatment day. Correlations between these measures will be determined between other cordance and total Hb levels obtained after the first week of treatment and MADRAS changes for the last day of treatment. Similar analyses will be conducted for changes in MADRAS scores between baseline and the follow-up visit.
Changes in MADRAS scores between baseline and the last treatment day | 6 Weeks
  The primary outcomes will be the correlations between EEG cordance or task-induced changes in frontal total Hb levels and changes in MADRAS scores between baseline and the last treatment day. Correlations between these measures will be determined between other cordance and total Hb levels obtained after the first week of treatment and MADRAS changes for the last day of treatment. Similar analyses will be conducted for changes in MADRAS scores between baseline and the follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ofra Sarid-Segal, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No